CLINICAL TRIAL: NCT05846503
Title: The Integrating HIV and hEART Health in South Africa Intervention Study
Brief Title: iHEART-SA Intervention Study
Acronym: iHEART-SA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Emory University (Other); Massachusetts General Hospital (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Professor Francois Venter, Executive Director, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: iHEART-SA IS
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; HIV
MeSH Terms: conditions — Hypertension | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Randomized cluster stepped-wedge study design where clinics will be assigned to a time at which they initiate the intervention. There are nine clinics which have been classification (low, medium and high) according to their volume. One clinic from each classification has been randomized to a cluster such that there are three clusters each with a low, medium and high volume clinic.
Masking Description: There is no masking. This is an intervention study without drugs. Intervention comprises training and education, data and feedback, and task shifting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Cluster of clinics receiving the five investigational interventions
  Interventions: Behavioral: 1. Quality and info management system
- Control (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: 1. Quality and info management system — 1. The intervention package prioritizes information and quality management with a focus on HTN screening, diagnosis, and treatment. From the point-of-care, flow charts placed in the patient file will ensure that vitals are performed in accordance with national guidelines.
  2. The care coordinator will present data to clinic staff in multi-disciplinary meetings, providing an opportunity for programmatic feedback and discussion.
  3. Patients will be encouraged to complete the vital signs measurements at each clinic visit. They will be provided with their BP readings and given info about what their reading means. They will be issued with pocket sized color coded booklets providing info on the measurement and what to do to control their BP.
  4. Task shifting: A care coordinator will be the champion of the intervention package for the clinic.
  5. All staff will receive apt training on how to use the patient flow chart, info management system and how to respond to abnormal BP values.
  Other Names: 2. Case review meetings; 3. Patient health education and support; 4. Task shifting; 5. HCW education and training
  Arms: Intervention

SUMMARY:
Using qualitative data during the formative phase the IHEART-SA research study filled deficiencies in knowledge regarding: 1) what barriers exist to integrating hypertension care within the HIV care setting in South Africa and, 2) how a hypertension care intervention can be adapted to effectively and sustainably function in this care setting. These data have been used to design a context-relevant intervention package for implementation in the next phase of effectiveness-implementation testing, answering the research question: How does an intervention aimed at enhancing hypertension diagnosis and management in people living with HIV improve the delivery of guideline-recommended care in primary healthcare clinics in Gauteng, South Africa, and hypertension control among patients?

The study will use an effectiveness-implementation study design. This design allows for the testing of strategies to promote integration of proven interventions in real-world practice (i.e., implementation strategies), while simultaneously assessing clinical effectiveness (i.e., patient level outcomes). For this the study will use a randomized cluster stepped-wedge study design where nine clinics (grouped in clusters of three) will be assigned to a time at which they initiate the intervention.

DETAILED DESCRIPTION:
Investigational interventions:

Implementation facilitation of improved hypertension screening and management in the HIV care setting through the iHEART-SA intervention model comprising:

1. Information management system
2. Task shifting
3. Audit and feedback
4. Healthcare worker education and training
5. Patient education and support

Study design:

Cluster randomized stepped wedge effectiveness-implementation type 2 hybrid

Study objectives:

1. Assess the short- and long-term effects of an implementation strategy (i.e., healthcare worker intervention) on the adoption and implementation of hypertension screening and treatment among healthcare workers
2. Assess the short- and long-term effects of a clinical intervention (i.e., patient-level intervention) on patient blood pressure control among patients living with HIV and hypertension

Duration of participation: 27 months Study duration: 37 months

Intervention audience:

1. Healthcare workers (nurses and doctors)
2. Adult patients living with HIV from the 9 primary healthcare clinics

ELIGIBILITY:
Inclusion Criteria:

Healthcare workers:

1. Adult >18 years men and women working in clinical roles at the selected clinics
2. Provide informed consent (only those participating in the qualitative components)

Patients:

1. Adults >18 years living with HIV and hypertension
2. Enrolled in the study clinic
3. Willing and able to provide informed consent

Exclusion Criteria:

Patients:

1. Unable or unwilling to provide informed consent
2. Planning to relocate or change service providers/clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4378 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Healthcare worker | 24 months
  Difference in percentage of patient visits with recorded BP measurement between intervention and control clinics
Patient | 12 months
  Difference in mean systolic BP between the intervention and control conditions

SECONDARY OUTCOMES:
Healthcare worker implementation | 24 months
  % of healthcare workers who implement the iHEART-SA package as intended at month 12 and month 24
Healthcare worker adoption | 24 months
  Participation rate and representativeness of healthcare workers who adopt the BP screening and treatment model
Healthcare worker maintenance - BP measurement | 12 months
  % of patients who had a BP measurement done at every clinic visit
Healthcare worker satisfaction | 24 months
  % of healthcare workers who are satisfied with all components of the intervention
Healthcare worker costing | 27 months
  Costs of each intervention components will be recorded as healthcare worker time, material costs, and healthcare/monitoring equipment
Patient adoption | 24 months
  Participation rate and representativeness of eligible patients who consent to chart review
Patient satisfaction | 24 months
  % of patients who are satisfied with all components of the intervention
Healthcare worker maintenance - BP management | 12 months
  % of patients who had an elevate BP managed at every visit post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Willem DF Venter, MD, PHD, Principal Investigator — Ezintsha, University of the Witwatersrand
Locations (1):
- Sunnyside Office Park, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galaviz KI, Patel SA, Siedner MJ, Goss CW, Gumede SB, Johnson LC, Ordonez CE, Laxy M, Klipstein-Grobusch K, Heine M, Masterson M, Mody A, Venter WDF, Marconi VC, Ali MK, Lalla-Edward ST. Integrating hypertension detection and management in HIV care in South Africa: protocol for a stepped-wedged cluster randomized effectiveness-implementation hybrid trial. Implement Sci Commun. 2024 Oct 14;5(1):115. doi: 10.1186/s43058-024-00640-6. PMID 39402688